CLINICAL TRIAL: NCT00007488
Title: Virologic Studies in Compartmental Samples From HIV-Infected Subjects Changing or Initiating Potent Antiretroviral Therapy
Brief Title: HIV in Specific Parts of the Body of Patients Who Are Changing or Starting Potent Anti-HIV Drugs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: A5077; AACTG A5077; ACTG A5077
Record Dates: First submitted 2000-12-23; First posted 2001-08-31 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Lymphoid Tissue; Viremia; RNA, Viral; Saliva; Anti-HIV Agents; Viral Load; Genitalia, Female; Genitalia, Male
MeSH Terms: conditions — HIV Infections; Viremia

SUMMARY:
The purpose of this study is to gain information on how the type and amount of HIV present in certain places in the body and in the blood are affected when potent (powerful) anti-HIV drugs are given.

Researchers know that the type and amount of HIV may differ in certain places in the body (called compartments) but are not sure how anti-HIV treatment affects these differences. This study gathers information to help understand how the virus grows and changes between blood and nonblood compartments in patients receiving anti-HIV treatment.

DETAILED DESCRIPTION:
The goal of antiretroviral therapy is maximal suppression of HIV-1 replication. Yet studies show that there is ongoing replication of latent virus in the blood and lymphoid tissues of some patients receiving potent antiretroviral therapy who have had suppressed plasma HIV-1 RNA levels for prolonged periods of time. This continued viral persistence and replication could eventually result in virologic failure and clinical progression as well as selection and transmission of resistant HIV-1. There is a need to identify, quantify, and determine significance of viral reservoirs in compartments other than blood. A5077 is designed to evaluate the relationship between viral load in blood and nonblood compartments and time to virologic failure in patients initiating or changing potent antiretroviral therapy.

Patients contribute samples of blood at study entry (prior to changing or initiating potent antiretroviral therapy), Week 8 and every 8 weeks thereafter until Week 96, and (if applicable) within 30 days of confirmed virologic failure. Samples of saliva and either genital secretions or lymphoid tissue, or both, are collected at study entry (prior to changing or initiating potent antiretroviral therapy), Weeks 16, 48, and 96, and within 30 days of confirmed virologic failure. Clinical assessments and medication updates are done at study visits. Blood samples are tested for HIV-1 genotypic resistance studies, HIV-1 proviral DNA studies, and HIV-1 quantitation. If total blood volumes exceed safe limits, blood samples will not be drawn for A5077 but the A5077 protocol team will request access to plasma and PBMC samples from any coenrolled study if applicable.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old.
* Are HIV-positive.
* Are changing or beginning anti-HIV therapy (not provided by the study). Anti-HIV therapy should be an approved 3-drug combination.
* Have a viral load of at least 2,000 copies/ml within 60 days of study entry.
* Have signed consent of parent or guardian if under 18 years of age.
* Are willing to contribute samples of blood, saliva, and either genital fluids or lymph tissue, or both, at study visits.
* Are willing to give permission to allow records from any coenrolled studies to be used while participating in this study.
* Have a negative pregnancy test within 14 days of study entry, if women able to have children. Women who become pregnant while on the study are allowed only to contribute blood and saliva samples until the pregnancy ends. After the pregnancy has ended, collection of genital fluids and/or lymphoid tissue will continue.
* Agree to receive HIV-related care at an AACTG site, if not enrolled in another AACTG trial.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have had any active opportunistic (AIDS-related) infection or disease, or have another illness occurring at the same time, or other infections, including an active lower genital tract infection that requires a new drug or change in drug in 14 days or less before study entry. There may be an exception for some conditions.
* Have used immunomodulatory agents in 14 days or less before study entry.
* Have had an immunization in 14 days or less before study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164
Dates: Start 2000-11; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejo Erice, Study Chair; Robert Coombs, Study Chair; Susan Fiscus, Study Chair
Locations (23):
- United States (23):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California, San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Univ of California San Francisco, San Francisco, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Emory Univ, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ of Minnesota, Minneapolis, Minnesota
  - Washington Univ / St Louis Connect Care, St Louis, Missouri
  - Washington Univ School of Medicine, St Louis, Missouri
  - Community Health Network Inc, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Derived] Kantor R, Bettendorf D, Bosch RJ, Mann M, Katzenstein D, Cu-Uvin S, D'Aquila R, Frenkel L, Fiscus S, Coombs R; ACTG A5077 Study Team. HIV-1 RNA levels and antiretroviral drug resistance in blood and non-blood compartments from HIV-1-infected men and women enrolled in AIDS clinical trials group study A5077. PLoS One. 2014 Apr 3;9(4):e93537. doi: 10.1371/journal.pone.0093537. eCollection 2014. PMID 24699474